CLINICAL TRIAL: NCT05882006
Title: A Multicenter Case-control Study of the Association Between the Presence of Gallstone Disease and Risk of Inflammatory Bowel Disease
Brief Title: Gallstones and Risk of Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Director of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: IBD Risk of Gallstones
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Gallstone; Crohn's disease; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Gallstones; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: IBD patients (including Crohn's disease and Ulcerative colitis)
  Interventions: Other: gallstones
- controls: Age, sex, and calendar-year matched controls sampled from non-IBD patients to be a round number of at least four times the number of cases
  Interventions: Other: gallstones

INTERVENTIONS:
Other: gallstones — fellow up if the patients have gallstones

SUMMARY:
The purpose of this study was to evaluate the association between gallstone disease and the risk of inflammatory bowel disease.

DETAILED DESCRIPTION:
Crohn's disease and ulcerative colitis , collectively known as inflammatory bowel diseases , have increased substantially over the past few decades affecting nearly 6.8 million individuals worldwide. The etiology of IBD remains obscure, possibly involving a complex interaction between the genetic, environmental or microbial factors and the immune responses. Gallstone disease is one of the most common and costly gastroenterological disorders, with a prevalence of 10-20% in Europe and America. Considering that gallstones and IBD also share specific risk factors, such as obesity, inappropriate diet and metabolic hormone levels, and have the pathophysiologic linkage, such as changes in gut microbiota composition and bile acid profile, the investigators propose that the occurrence of gallstones may predict the subsequence risk of IBD. However, investigations concerning the association is lacking.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years old
* IBD established by standard criteria, either Crohn's disease or ulcerative colitis

Exclusion Criteria:

* Pregnant or nursing woman;
* Prior abdominal surgery related to IBD, such as subtotal or total colectomy;
* HIV infection or any congenital immunodeficiency at the time of inclusion;
* Post organ transplant patients;
* Patients suffering from cancer currently or in the past;
* Patients suffering from significant cardiovascular disease;
* Patients suffering from significant respiratory diseases;
* Patients suffering from any other chronic severe diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IBD patients
Sampling Method: Probability Sample
Enrollment: 5035 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
The prevalence of gallstone disease among patients with or without IBD | 10 years
  We assess the prevalence as the number of gallstone diseases divided by the number of IBD patients or non-IBD patients. Gallstone disease was diagnosed as presence of gallstones, cholecystectomy, choledocholithotomy and Endoscopic Retrograde Cholangio-Pancreatography (ERCP).
The odds ratio of the association between the presence of gallstone disease and risk of inflammatory bowel disease | 10 years
  The odds ratio is a ratio of two sets of odds: the odds in case group (gallstone diseases with IBD divided by non-gallstone disease with IBD) versus the odds in control group (gallstone diseases without IBD divided by non-gallstone disease without IBD). Finally, we can calculate the odds ratio by dividing the ratio of the case group by the ratio of the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D., Study Chair — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (4):
- China (4):
  - Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Wuwei Tumor Hospital, Wuwei, Gansu
  - The Seventh Affiliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
After completed

REFERENCES:
- [Background] GBD 2017 Inflammatory Bowel Disease Collaborators. The global, regional, and national burden of inflammatory bowel disease in 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet Gastroenterol Hepatol. 2020 Jan;5(1):17-30. doi: 10.1016/S2468-1253(19)30333-4. Epub 2019 Oct 21. PMID 31648971
- [Background] Lammert F, Gurusamy K, Ko CW, Miquel JF, Mendez-Sanchez N, Portincasa P, van Erpecum KJ, van Laarhoven CJ, Wang DQ. Gallstones. Nat Rev Dis Primers. 2016 Apr 28;2:16024. doi: 10.1038/nrdp.2016.24. PMID 27121416
- [Derived] Mi N, Yang M, Wei L, Nie P, Zhan S, Nguyen LH, Smith FG, Acharjee A, Liu X, Huang J, Xia B, Yuan J, Meng W. Gallstone Disease Is Associated With an Increased Risk of Inflammatory Bowel Disease: Results From 3 Prospective Cohort Studies. Am J Gastroenterol. 2025 Jan 1;120(1):204-212. doi: 10.14309/ajg.0000000000003111. Epub 2024 Oct 4. PMID 39364876